CLINICAL TRIAL: NCT04066101
Title: Variants in Taste Genes on Caries Risk and Caries Activity Status
Brief Title: TAS1R1, TAS1R3, TLR2, TLR4, CA6 Gene Polymorphism on Dental Caries
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gul Yildiz Telatar, Principal Investigator, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2016/30
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: High Caries Risk; Low Caries Risk
Keywords: caries risk, gene polymorphisms
MeSH Terms: interventions — Genotype; Dental Caries Activity Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA for genetic analysis was isolated from buccal epithelial cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high caries risk: 100 adults will be allowed in the high caries risk group according to DMFT index (DMFT ≥ 14)
  Interventions: Genetic: high caries risk; Other: caries activity
- low caries risk: 100 adults will be allowed in the low caries risk group according to DMFT index (DMFT ≤ 5)
  Interventions: Genetic: high caries risk; Other: caries activity

INTERVENTIONS:
Genetic: high caries risk — DNAs were obtained from epithelial cells in buccal mucosa and were extracted with Genomic DNA Isolation Kit Genotyping for a variant was carried out on a Roche Applied Science LightCycler® 480 (Roche Diagnostics GmbH, Mannheim, Germany) with real-time polymerase reaction of Taqman
  Other Names: DNA isolation, genotyping
Other: caries activity — Dental caries lesions of all patient scored as initial, moderate or advanced caries
  Initial lesion; clinically detectable lesion Moderate; visible signs of enamel breakdown Advanced; enamel was fully cavitaed

SUMMARY:
The aim of this study is to examine the effects of TAS1R1, TAS1R3, TLR2, TLR4, CA6, gene polymorphism on caries risk in adults.

DETAILED DESCRIPTION:
To date, genes can be grouped into categories based on the factor influencing dental caries. The major candidate gene categories to date include enamel formation genes, immune response genes, genes related to saliva, and genes related to taste and dietary habits.

CA6 exists in the human saliva and has a critical role of buffering, immune response and taste.Toll-like receptors are expressed in the tongue gustatory papillae where they may initiate immune responses to pathogens.Genetic variations in the TAS1R1 and TAS1R3 for umami cause perception of these tastes differently.

ELIGIBILITY:
Inclusion Criteria:

* adult be between 25 and 44 years old
* subject has DMFT (Decayed, Missing, Filled, Permanent Tooth) ≥ 5, or, DMFT ≥14
* same oral health, diet and socioeconomic status

Exclusion Criteria:

* systemic or genetic disorders
* orthodontic appliances
* pregnant women

Ages: 25 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Power analysis was performed with the G-Power software package. It was determined that a total of 200 patients will be needed: 100 (DMFT ≤ 5) for the low caries risk group and 100 (DMFT ≥ 14) for the high caries risk group
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Past caries experience | 4 months
  Each tooth will be examined and recorded as decayed, missing, or filled (DMFT). Caries will be defined in accordance with the World Health Organization (WHO 1997) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Gül Yıldız Telatar, Dr., Principal Investigator — Recep Tayyip Erdogan University Dentistry Faculty
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be available within 6 months of study completion

REFERENCES:
- [Background] Yildiz G, Ermis RB, Calapoglu NS, Celik EU, Turel GY. Gene-environment Interactions in the Etiology of Dental Caries. J Dent Res. 2016 Jan;95(1):74-9. doi: 10.1177/0022034515605281. Epub 2015 Sep 16. PMID 26377569
- [Derived] Yildiz Telatar G, Saydam F, Guzel AI, Telatar BC. Variants in taste genes on caries risk and caries activity status. Med Mol Morphol. 2020 Dec;53(4):244-251. doi: 10.1007/s00795-020-00263-5. Epub 2020 Aug 7. PMID 32770263
- See also: Gene-environment Interactions in the Etiology of Dental Caries. — http://www.ncbi.nlm.nih.gov/pubmed/26377569